CLINICAL TRIAL: NCT02374736
Title: A Pilot Study on the Effect of Privigen Against Graft Loss: Interventional Study of Kidney Transplant Recipients at Risk for Graft Loss Through Antibody-mediated Rejection
Brief Title: Effect of Privigen Against Graft Loss
Acronym: InAuGuRAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CSL Behring (Industry); Association ASLUMARE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140501; 2014-003707-30 (EudraCT Number)
Record Dates: First submitted 2015-01-20; First posted 2015-03-02 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Kidney Transplantation
Keywords: recipients; Subclinical Antibody-mediated rejection (ABMR); Intravenous immunoglobulins (IVIg); Donor-specific antibodies (DSA)
MeSH Terms: interventions — Immunoglobulins, Intravenous; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human normal immunoglobulin G (IgG > 98 % purity) (Experimental): All subjects will be treated for 6 months. The treatment will start the day of inclusion (M0).
  Privigen will be given as 2 g/kg for 2 days/month. The maximum daily dose authorized will be 80g.
  The infusion rates are the recommended rates for Privigen in other indications and are in line with the market authorization for Privigen:
  * Infusions should start at a rate of 0.5 mg/kg/min (0.005 mL/kg/min; 0.3 mL/kg/h; 30 mg/kg/h). If well tolerated within 30 min, the rate can be increased in a first step to 1.0 mg/kg/min (0.01 mL/kg/min; 0.6 mL/kg/h; 60 mg/kg/h) for another 30 min.
  * If well tolerated, a stepwise increase to a maximum of 8 mg/kg/min (0.08 mL/kg/min; 4.8 mL/kg/h; 480 mg/kg/h) is allowed at the discretion of the investigator.
  Interventions: Drug: Privigen (Human normal immunoglobulin G (IgG > 98 % purity))

INTERVENTIONS:
Drug: Privigen (Human normal immunoglobulin G (IgG > 98 % purity)) — Privigen (CSL Behring AG, Bern, Switzerland) 10% liquid human IgG for intravenous administration, 2 g/kg, given as 2 g/kg for 2 days/month for 6 months (maximum dose: 80 g/day).
  Privigen will be provided in vials containing 10 g IgG in 100 mL.

SUMMARY:
The principal objective of this pilot study is to determine whether the progression of chronic antibody-mediated rejection (ABMR) could be minimized by the post-transplant administration of high dose of Intravenous Immunoglobulins (IVIg).

We test the hypothesis that repetitive IVIg administration reduces or stabilize the progressive loss of transplant function and the evolution to chronic ABMR in stable kidney transplant patients with HLA-DSA developed post-transplantion (de novo HLA-DSA) and concomitant humoral graft injury.

DETAILED DESCRIPTION:
The aim of this study is to assess the effect of IVIg associated to conventional immunosuppressive treatment in 15 stable transplant recipients with post-transplant de novo HLA-DSA and histological humoral lesions.

The study will include 2 periods:

* Treatment period,
* Follow-up period. The treatment will start the day of inclusion (M0): Privigen will be given as 2 g/kg for 2 days/month for 6 months (maximum dose: 80 g/day).

Evaluation at the end of treatment will take place on month 6 (M6). Evaluation at the end of follow up will take place on month 12 (M12).

Blood and urine samples will be collected on day of inclusion (M0), before each infusion of Privigen, at M6 and M12 for biological analysis (serum creatinine, glomerular filtration rate, proteinuria).

Blood samples will be collected on day of inclusion (M0), at M6 and M12 for immunoassay (HLA-DSA mean fluorescence intensity).

Blood sample will be collected on day of inclusion (M0) to provide a DNA bank. Blood samples will be collected on day of inclusion (M0), before each infusion of Privigen and at M6 for IgG dosage.

Blood samples will be collected on day of inclusion (M0), before each infusion of Privigen, at M6 and M12 to provide a serum bank.

Blood samples will be collected on day of inclusion (M0), before each infusion of Privigen, at M6 and M12 for haematology, blood chemistry and Coombs test.

Histological characteristics (kidney biopsies) will be performed on M0 and M6. The M6 biopsy is specifically requested by the protocol and differs from the usual practice, where it is usually performed at M12 post transplantation.

Infectious and clinical events (deceased patients, graft loss, acute biopsy-proven rejection episode and infectious diseases) will be recorded during the follow-up period.

Histology of for-cause biopsies will be performed according to center practice. We recommend a graft biopsy for patients with acute allograft dysfunction (20% increase of creatinine) without current evident causes of graft dysfunction.

The maximum study duration for a subject, between inclusion and follow-up visits, will be 12 months and the estimated length of time needed to complete the entire study (from enrolment of the first subject to completion of the last subject) 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Deceased donor kidney transplant recipients between 3 and 12 months post transplantation.
2. At least 18 years old.
3. With stable renal function assessed within 30 days before inclusion and with delta GFR (MDRD) lower than 10 ml/min (latest result versus the average of the two previous values).
4. Presence of at least one circulating HLA-DSA class I or II against HLA-A, -B, -DR, -DQ, -DP, -C (MFI ≥ 1000) as assessed by Luminex single antigen technique within 30 days before inclusion.
5. With histological markers of active antibody-mediated injury as defined by the microcirculation inflammation score (g, ptc scores defined by current Banff criteria) on protocol biopsies performed at M3 or M12 post-transplantation, or if required between three and twelve months post transplantation (1 ≤ g+ptc ≤ 3).
6. Able to comply with the study procedures and follow the study instructions.
7. Who have read the information sheet and signed the informed consent form.

Exclusion Criteria:

1. Acute renal dysfunction at the time of enrolment: decrease of GFR higher or equal to 10 ml/min (latest result versus the average of the two previous values), or 20% increase of serum creatinine.
2. Previous episode of ABMR.
3. Previous treatment with plasmapheresis, IVIg, within 2 months prior to inclusion

3b. Previous treatment with rituximab, eculizumab or bortezomib within 1 year prior to inclusion

4. Major lesions of active antibody-mediated injury, as defined by Banff criteria, such as g + ptc >3 or chronic transplant glomerulopathy (cg>0).

5. History of cardiac insufficiency (New York Heart Association [NYHA] III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease, congestive heart failure or severe hypertension.

6. History of thrombotic episodes (deep vein thrombosis, myocardial infarction, cerebrovascular accident).

7. Known allergic or other severe reactions to blood products including intolerability to previous IVIg (i.e. severe headache, hypersensitivity, intravascular hemolysis).

8. Subject with a known deficit in IgA, with antibodies against IgA. 9. Known hyperprolinemia.

10. Ongoing HIV, hepatitis C and hepatitis B infection.

11. Any condition (including alcohol, drug or medication abuse) that is likely to interfere with evaluation of the study product or satisfactory conduct of the study.

12. Not able to comply with study procedures and treatment regimen.

13. Pregnant or lactating women or women of childbearing potential without effective method of contraception (oral contraceptive pill, intra-uterine contraceptive device, contraceptive implant or condom).

14. Participation in any other study involving investigational products, concomitantly or within 30 days prior to entry in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Graft function: estimation of change from baseline Glomerular Filtration Rate (GFR) using MDRD | at months 6
  using Modification of Diet in Renal Disease (MDRD) equation at M6
Graft function: estimation of change from baseline Glomerular Filtration Rate (GFR) using MDRD | at months 12
  using Modification of Diet in Renal Disease (MDRD) equation at M12

SECONDARY OUTCOMES:
Change of proteinuria from baseline | months 6 and months 12
  Change of proteinuria value at M6 and M12 compared to M0. The proteinuria is measured from blood sample
Change of HLA-DSA from baseline | months 6 and months 12
  The presence of HLA-DSA will be analyzed using Luminex single-antigen assays at M6 and M12 compared to M0. The HLA-DSA is measured from blood sample
Change of Histological characteristics from baseline | at months 6
  A kidney biopsy will be performed at M6 and compared to M0
IgG dosage | up to months 6
  IgG dosage will be performed at M0, before each Privigen infusion and at M6
Infectious events reported during the study period | up to months 12
  Infectious events will be reported from M0 to M12.

CONTACTS AND LOCATIONS:
Overall Officials: Denis GLOTZ, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Néphrologie et transplantation rénale - HU Saint-Louis, Paris, Île-de-France Region, France